CLINICAL TRIAL: NCT02341391
Title: A Dose-escalating, Single-center, Phase I Clinical Trial to Investigate the Safety and Biological Efficacy of TissueGene-C in Degenerative Arthritis Patients.
Brief Title: Safety and Biological Efficacy Study of TisssueGene-C to Degenerative Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kolon Life Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TGC-KI-01
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Degenerative Arthritis
Keywords: chondrocyte cells; Osteoarthritis; gene therapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TissueGene-C(Low dose) (Experimental): Single intra-articular injection to the damaged knee joint at doses of 3.0 x 10^6 cells
  Interventions: Biological: TissueGene-C(Low dose)
- TissueGene-C(Medium dose) (Experimental): Single intra-articular injection to the damaged knee joint at doses of 1.0 x 10^7 cells
  Interventions: Biological: TissueGene-C(Medium dose)
- TissueGene-C(High dose) (Experimental): Single intra-articular injection to the damaged knee joint at doses of 3.0 x 10^7 cells
  Interventions: Biological: TissueGene-C(High dose)

INTERVENTIONS:
Biological: TissueGene-C(Low dose) — 3.0 x 10^6 cells
  Arms: TissueGene-C(Low dose)
Biological: TissueGene-C(Medium dose) — 1.0 x 10^7 cells
  Arms: TissueGene-C(Medium dose)
Biological: TissueGene-C(High dose) — 3.0 x 10^7 cells
  Arms: TissueGene-C(High dose)

SUMMARY:
The primary purpose of the this study is to evaluate the safety of TissueGene-C, a gene therapy product that uses allogenic human chondrocytes expressing Transforming Growth Factor(TGF)-β1 by assessing the inflammation at the injection site, the incidence and severity of the adverse events, the physical examination findings, and the laboratory test results after the intra-articular injection of TissueGene-C.

And Secondary purpose is to evaluate the biological efficacy (knee pain, range of motion, functional tests, and MRI) of TissueGene-C and the distribution of TissueGene-C outside the injection site.

DETAILED DESCRIPTION:
TissueGene-C is a biological new drug which consists of normal chondrocyte cells and transduced chondrocyte cells that express growth factor to modify osteoarthritis symptom for long term period.

During clinical trial Phase 1, we compare three different dose levels of TisssueGene-C in 6 months with 12 outpatients with degenerative arthritis. The patients are randomized by three different dose levels of TisssueGene-C in 1:1:1 ratio, and they are monitored and recorded for alleviating symptoms, sports activities, function of the knee, and the presence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients
2. Patients aged 45 years or more with Grade IV [based on the International Cartilage Repair Society(ICRS) evaluation criteria from the MRI scan results] degenerative arthritis of the knee, whose symptoms had not been relieved by the conventional symptomatic treatment
3. Healthy, with no major physical examination, hematology, serum chemistry, and urine test findings and no significant medical history
4. Patients with cartilage damage sized 2-6 cm2 (based on the ICRS evaluation criteria from the MRI scan results)
5. Voluntarily agreed to participate in this study and signed the informed consent form

Exclusion Criteria:

1. Showed clinically significant hematology, serum chemistry, or urine test results at the screening visit
2. Took an anti-inflammatory medication (prescribed or over-the-counter), including natural medicine, within 14 days from the administration of the investigational product
3. Has a history of drug abuse within one year from the enrollment, or the urine test or blood alcohol test result was positive at the screening visit
4. Received any injection in the target knee within two months before the initiation of the study
5. Pregnant or breastfeeding female
6. With another joint disease apart from degenerative arthritis (e.g., systemic rheumatic inflammatory disease associated with the knee or chondrocalcinosis, hemachromatosis, inflammatory arthritis, necrosis of the trochanter, Paget's disease adjacent to a joint in the femur or the tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's disease in the knee joint, villonodular synovitis, and synovial chondromas)
7. With an infectious disease, including HIV or hepatitis (HBV/HCV)
8. With a history any of the following clinically significant diseases:

   * heart disease [e.g., myocardial infarction, arrhythmia, other serious heart disease, coronary artery bypass graft (CABG)]
   * kidney disease (e.g., chronic renal failure, glomerulonephritis)
   * liver disease (e.g., liver cirrhosis, fatty liver, acute or chronic liver disease)
   * endocrine disease (e.g., hyperthyroidism, hypothyroidism, thyroiditis, diabetes insipidus, Cushing's disease)
   * insulin-dependent diabetes mellitus
   * medical history of or current malignant tumor In particular, the tumors that TissueGene-C may aggravate can be screened using the following tests

     * Leukemia : White Blood Cell level in the hematology
     * Osteochondroma, Chondromas, Chondroblastoma, Chondromyxoid fibroma, Chondrosarcoma : Alkaline phosphatase level in the hematology
9. Participated in another clinical trial (using the investigational drug or a medical device) within 30 days before enrollment in this study
10. Showed positive drug test results at the screening visit
11. Did not agree to use a contraceptive method (male and female)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events after the administration of TissueGene-C | 6 months
  Number of Participants with Adverse Events after the administration of TissueGene-C

SECONDARY OUTCOMES:
Changes in MRI scan | before and 28 days, 3 months, and 6 months
  Change in the MRI scan results after the administration of TissueGene-C
Change in the Knee Society Clinical Rating System(KSCRS) test results | before and 7 days, 14 days, 21 days, 28 days, 3 months, and 6 months
  Comparative Evaluation of knee exam
Changes in WOMAC scores | before and 7 days, 14 days, 21 days, 28 days, 3 months, and 6 months
  Pain, stiffness, and physical function of the knee will be measured by the Western Ontario and McMaster Universities(WOMAC)
Changes in 100 mm-VAS | before and 7 days, 14 days, 21 days, 28 days, 3 months, and 6 months
  Pain of the knee will be measured by the 100mm Visual Analogue Scale (VAS)
Analysis of the TGF-β1 expression using Enzyme-linked Immunosorbent Assay(ELISA) and Polymerase Chain Reaction(PCR) | before and 7 days, 14 days, 21 days, 28 days, 3 months, and 6 months
  Analysis of the TGF-β1 expression using Enzyme-linked Immunosorbent Assay(ELISA) and Polymerase Chain Reaction(PCR)
Replication-competent retrovirus test (RCR test) | before and 7 days, 14 days, 21 days, 28 days, 3 months, and 6 months
  Replication-competent retrovirus test (RCR test)

CONTACTS AND LOCATIONS:
Overall Officials: Chul Won Ha, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea